CLINICAL TRIAL: NCT01081522
Title: A Preliminary, Non-comparative Study to Evaluate a Bioresorbable Wound Scaffold in Acute Wounds
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Dheerendra Kommala, MD, Convatec Inc.
Other Study IDs: CW-0510-09-U352
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue (3mm punch biopsy)

SUMMARY:
As this is a proof-of-concept study, the primary objective is to provide preliminary data on the safety and efficacy of Bioresorbable Wound Scaffold in the management of acute wounds left to heal by secondary intent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent.
* Subjects who have an excised pilonidal sinus wound left to heal by secondary intent.
* Subjects who are willing to commit to having two biopsies being taken during the study.

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product
* Subjects whose wound is infected
* Subjects who have participated in a previous clinical study within the past 3 months
* Subjects' with a known history of poor compliance with medical treatments
* Subjects who are pregnant (where pregnancy is a possibility, a pregnancy testing kit will be provided)
* Necrotic/sloughy wounds unless surgically debrided prior to enrolment
* Medical or emotional risk associated with the potential biopsy that outweighs the risk of not taking a biopsy as determined by the investigator
* Subjects exhibiting any other medical condition which, according to the Investigator, justifies the subject's exclusion from the study
* Subjects with impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dheerendra Kommala, MD, Study Director — ConvaTec Inc.
Locations (3):
- Hillerod Hospital, Hillerød, Dk 3400, Denmark
- United Kingdom (2):
  - Wound Healing Research Unit, Heathpark, Cardiff
  - Scunthorpe General Hospital, Scunthorpe, North Lincolnshire